CLINICAL TRIAL: NCT03988075
Title: Use of Enhanced Recovery After Surgery (ERAS) in Minimizing Opioid Use for Patients Undergoing Thyroidectomy
Brief Title: Non-opioid Based Pain Control After Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-022
Record Dates: First submitted 2019-05-14; First posted 2019-06-17 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pain; Thyroidectomy
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomized to one of two study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetaminophen and hydrocodone based pain control (Active Comparator): Patients receive acetaminophen 650mg every 4 for pain level 1-3, hydrocodone/acetaminophen 5/325mg every 4 for pain level 4-6, or hydrocodone/acetaminophen 10/650mg every 4 for pain level 7-10 on as needed basis.
  Interventions: Other: Acetaminophen and hydrocodone based pain control
- Acetaminophen and ibuprofen based pain control (Experimental): Patients receive standing dose of acetaminophen 650mg every 8 hours and ibuprofen 800mg every 8 hours with alternating ibuprofen and acetaminophen every 4 hours.
  Interventions: Other: Acetaminophen and ibuprofen based pain control

INTERVENTIONS:
Other: Acetaminophen and hydrocodone based pain control — Patients receive acetaminophen 650mg every 4 for pain level 1-3, hydrocodone/acetaminophen 5/325mg every 4 for pain level 4-6, or hydrocodone/acetaminophen 10/650mg every 4 for pain level 7-10 on as needed basis.
  Arms: Acetaminophen and hydrocodone based pain control
Other: Acetaminophen and ibuprofen based pain control — Patients receive standing dose of acetaminophen 650mg every 8 hours and ibuprofen 800mg every 8 hours with alternating ibuprofen and acetaminophen every 4 hours.
  Arms: Acetaminophen and ibuprofen based pain control

SUMMARY:
Pain control modalities were evaluated after thyroidectomy.

DETAILED DESCRIPTION:
Pain control modalities were evaluated after thyroidectomy. Patients were randomized to one of two pain control regimens. The control group received conventional opioid based post operative analgesia while the test group received an enhanced recovery after surgery (ERAS) based anesthesia with use of acetaminophen and non-steroidal anti-inflammatory drugs for the post operative period with opioid medications available for break through pain only. Pain scores (measured on visual analog scale) and opioid use (measured in morphine equivalent dose) were measured after completion of the operation.

ELIGIBILITY:
Inclusion Criteria:

* thyroid disease

Exclusion Criteria:

* currently on opioid pain medications
* on opioid pain meds in last 30 days
* cannot take non-opioid medications
* require more extensive operation than thyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale pain level | 1 hour post operatively
  Pain level from 0 (no pain) to 10 (worst pain imaginable).
visual analog scale pain level | 6 hour post operatively
  Pain level from 0 (no pain) to 10 (worst pain imaginable).
visual analog scale pain level | 24 hour post operatively
  Pain level from 0 (no pain) to 10 (worst pain imaginable).
visual analog scale pain level | 7 days post operatively
  Pain level from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
opioid use | with the first 24 hours post operatively
  the dose of opioid received by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Erin Felger, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Francis DO, Randolph G, Davies L. Nationwide Variation in Rates of Thyroidectomy Among US Medicare Beneficiaries. JAMA Otolaryngol Head Neck Surg. 2017 Nov 1;143(11):1122-1125. doi: 10.1001/jamaoto.2017.1746. PMID 29049468
- [Result] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Result] Wilmore DW, Kehlet H. Management of patients in fast track surgery. BMJ. 2001 Feb 24;322(7284):473-6. doi: 10.1136/bmj.322.7284.473. No abstract available. PMID 11222424
- [Result] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591